CLINICAL TRIAL: NCT03226119
Title: HTLV Blot 2.4 Post-Market Clinical Study of Neurological Disorders and HTLV Positive Specimens
Brief Title: MP Diagnostics HTLV Blot 2.4 Post-Market Clinical Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MP Biomedicals, LLC (Industry)
Collaborators: MP Biomedicals Asia Pacific Pte. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MP-EIA-HTLV-002B
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2017-09

CONDITIONS: HTLV-I Infections; HTLV-II Infections; Human T-lymphotropic Virus 1; Human T-lymphotropic Virus 2; HTLV I Associated T Cell Leukemia Lymphoma; HTLV I Associated Myelopathies
Keywords: HTLV; Confirmatory; Supplemental; Blot; HTLV-I; HTLV-II
MeSH Terms: conditions — HTLV-I Infections; HTLV-II Infections; Leukemia-Lymphoma, Adult T-Cell; Paraparesis, Tropical Spastic

STUDY DESIGN:
Intervention Model Description: Cohort A: 100 Neurological Disorder Specimens Cohort B: 50 HTLV Known Positive Specimens
Who Masked: Investigator
Masking Description: Clinical Sites and the Reference Core-Lab will be masked of specimen disease state
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- HTLV Infected (n=50) (Experimental): Serum/plasma specimens which are HTLV I, HTLV II or HTLV I/II known positive (KP)
  Interventions: Diagnostic Test: MP Diagnostics HTLV Blot 2.4
- Neurological Disorders (n=100) (Experimental): Serum/plasma specimens with symptoms or any of the following neurological disorders: Acute Disseminated Encephalitis, Amyotrophic Lateral Sclerosis, Autonomic Dysfunction, Conus Medularis Syndrome, Chronic Inflammatory Demyelinating Polyneuropathy (CIDP), Dermatomyositis, HAM-TSP, Meningitis, Mild Cognitive Impairment, Multiple Sclerosis, Polymyositis, Spastic Paraparesis, Sciatica
  Interventions: Diagnostic Test: MP Diagnostics HTLV Blot 2.4

INTERVENTIONS:
Diagnostic Test: MP Diagnostics HTLV Blot 2.4 — HTLV I/II Confirmation and Differentiation
  Other Names: HTLV I/II Western Blot Assay

SUMMARY:
This post-market study is intended to assess the performance of the HTLV Blot 2.4 in repository serum/plasma specimens with neurological disorders (n=100) or an HTLV known positive infection (n=50).

DETAILED DESCRIPTION:
The HTLV Blot 2.4 Post-Market Clinical Study is an open-label, multi-center, single-blind clinical study of neurological disorders (n=100) and HTLV known-positive (KP) specimens (n=50). This study is being conducted to support additional labeling claims and to further assess the sensitivity and specificity of the HTLV Blot 2.4 in specimens with neurological disorders and HTLV known positive specimens.

ELIGIBILITY:
Inclusion Criteria:

All Specimens:

* Male or female
* Biorepository specimen de-identified of PHI
* Specimen meets HTLV Blot 2.4 labeling collection/handling criteria

HTLV Positive Specimens:

Specimens with a known positive infection of HTLV I, HTLV II or HTLV I/II

Neurological Disorders:

Specimens with a diagnosis or symptoms consistent with any of the following neurological disorders:

* Acute Disseminated Encephalitis
* Amyotrophic Lateral Sclerosis (ALS)
* Autonomic Dysfunction
* Conus Medularis Syndrome
* Chronic Inflammatory Demyelinating Polyneuropathy
* Dermatomyositis
* HTLV associated myelopathy-tropical spastic paraparesis (HAM-TSP)
* Meningitis
* Mild Cognitive Impairment
* Multiple Sclerosis (MS)
* Polymyositis
* Spastic Paraparesis
* Sciatica

Exclusion Criteria:

HTLV Infected:

* specimens with a known infection or history of HIV, HCV or HBV
* specimens not meeting specimen labeling collection / handling criteria

Neurological Disorders

* specimens not meeting specimen labeling collection / handling criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
To demonstrate ≥95% agreement of HTLV Blot 2.4 results with the Reference Core Laboratory HTLV Algorithm in 100 Neurological Disorder Specimens | 3 months
To demonstrate HTLV Blot 2.4 sensitivity of ≥97.5% in 50 HTLV Known Positive Specimens | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sara Dionne, PhD, Principal Investigator — LABS, Inc.
Locations (3):
- United States (3):
  - LABS, Inc., Philadelphia, Pennsylvania
  - Qualtex Laboratories, San Antonio, Texas
  - Eastern Virginia Medical School (EVMS), Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
All clinical study data will be compiled and shared with investigators following database lock.
Supporting Information: Study Protocol, CSR
Time Frame: Q4 2017

REFERENCES:
- [Background] Miller L. Profile of the MP Diagnostics HTLV Blot 2.4 test: a supplemental assay for the confirmation and differentiation of antibodies to HTLV-1 and HTLV-2. Expert Rev Mol Diagn. 2016;16(2):135-45. doi: 10.1586/14737159.2016.1123622. Epub 2016 Jan 11. PMID 26589659